CLINICAL TRIAL: NCT04553692
Title: An Open-label, Multicenter, Phase 1a/1b Study of Aplitibart (IGM-8444) As a Single Agent and in Combination in Participants with Relapsed, Refractory, or Newly Diagnosed Cancers
Brief Title: Phase 1a/1b Study of Aplitabart (IGM-8444) Alone or in Combination in Participants with Relapsed, Refractory, or Newly Diagnosed Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due strategic corporate pivot to focus on auto-immune indications
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IGM-8444-001
Record Dates: First submitted 2020-09-04; First posted 2020-09-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor; Colorectal Cancer; Non Hodgkin Lymphoma; Sarcoma; Chondrosarcoma; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia; Acute Myeloid Leukemia
Keywords: Relapsed and/or Refractory; Metastatic Cancer; Advanced Tumors; Hematological cancer; Newly diagnosed
MeSH Terms: conditions — Colorectal Neoplasms; Lymphoma, Non-Hodgkin; Sarcoma; Chondrosarcoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Neoplasm Metastasis | interventions — IFL protocol; Fluorouracil; Leucovorin; Irinotecan; Bevacizumab; birinapant; venetoclax; Gemcitabine; Docetaxel; Azacitidine

STUDY DESIGN:
Masking Description: Phase 1a is non-randomized; Ph1b is randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Ph1a: Aplitabart Single Agent Alternate Dosing Escalation (Experimental): Aplitabart will be administered intravenously as a single agent on an alternate dosing schedule.
  Interventions: Drug: Aplitabart (IGM-8444)
- Ph1a: Aplitabart + FOLFIRI ± bevacizumab Escalation and Expansion (Experimental): Aplitabart will be administered intravenously in combination with FOLFIRI± bevacizumab.
  Interventions: Drug: Aplitabart (IGM-8444); Drug: FOLFIRI; Drug: Bevacizumab (and approved biosimilars)
- Ph1a: Aplitabart + Birinapant Escalation and Expansion (Experimental): Aplitabart will be administered intravenously in combination with Birinapant which will also be administered intravenously.
  Interventions: Drug: Aplitabart (IGM-8444); Drug: Birinapant
- Ph1a: Aplitabart + Venetoclax Escalation and Expansion (Experimental): Aplitabart will be administered intravenously in combination with Venetoclax.
  Interventions: Drug: Aplitabart (IGM-8444); Drug: Venetoclax
- Ph1a: Aplitabart + Docetaxel + Gemcitabine Escalation and Expansion (Experimental): Aplitabart will be administered intravenously in combination with Docetaxel and Gemcitabine.
  Interventions: Drug: Aplitabart (IGM-8444); Drug: Gemcitabine; Drug: Docetaxel
- Ph1a: Aplitabart + Venetoclax + Azacitidine Escalation and Expansion (Experimental): Aplitabart will be administered intravenously in combination with Venetoclax and Azacitidine.
  Interventions: Drug: Aplitabart (IGM-8444); Drug: Venetoclax; Drug: Azacitidine
- Ph1b: Aplitabart + FOLFIRI + Bevacizumab (Experimental): Aplitabart will be administered intravenously in combination with FOLFIRI + bevacizumab
  Interventions: Drug: Aplitabart (IGM-8444); Drug: FOLFIRI; Drug: Bevacizumab (and approved biosimilars)
- Ph1b: FOLFIRI + Bevacizumab (Experimental): Standard of Care FOLFIRI + bevacizumab will be administered intravenously
  Interventions: Drug: FOLFIRI; Drug: Bevacizumab (and approved biosimilars)

INTERVENTIONS:
Drug: Aplitabart (IGM-8444) — DR5 Agonist Investigational Drug
  Arms: Ph1a: Aplitabart + Birinapant Escalation and Expansion; Ph1a: Aplitabart + Docetaxel + Gemcitabine Escalation and Expansion; Ph1a: Aplitabart + FOLFIRI ± bevacizumab Escalation and Expansion; Ph1a: Aplitabart + Venetoclax + Azacitidine Escalation and Expansion; Ph1a: Aplitabart + Venetoclax Escalation and Expansion; Ph1a: Aplitabart Single Agent Alternate Dosing Escalation; Ph1b: Aplitabart + FOLFIRI + Bevacizumab
Drug: FOLFIRI — Chemotherapy Regimen
  Other Names: Fluorouracil or 5-FU; Leucovorin; Irinotecan
  Arms: Ph1a: Aplitabart + FOLFIRI ± bevacizumab Escalation and Expansion; Ph1b: Aplitabart + FOLFIRI + Bevacizumab; Ph1b: FOLFIRI + Bevacizumab
Drug: Bevacizumab (and approved biosimilars) — Targeted Therapy
  Other Names: Avastin
  Arms: Ph1a: Aplitabart + FOLFIRI ± bevacizumab Escalation and Expansion; Ph1b: Aplitabart + FOLFIRI + Bevacizumab; Ph1b: FOLFIRI + Bevacizumab
Drug: Birinapant — SMAC-mimetic Investigational Drug
  Arms: Ph1a: Aplitabart + Birinapant Escalation and Expansion
Drug: Venetoclax — Targeted Therapy
  Other Names: Venclexta
  Arms: Ph1a: Aplitabart + Venetoclax + Azacitidine Escalation and Expansion; Ph1a: Aplitabart + Venetoclax Escalation and Expansion
Drug: Gemcitabine — Chemotherapy
  Other Names: Gemzar
  Arms: Ph1a: Aplitabart + Docetaxel + Gemcitabine Escalation and Expansion
Drug: Docetaxel — Chemotherapy
  Other Names: Taxotere; Docefrez
  Arms: Ph1a: Aplitabart + Docetaxel + Gemcitabine Escalation and Expansion
Drug: Azacitidine — Chemotherapy
  Other Names: VIDAZA
  Arms: Ph1a: Aplitabart + Venetoclax + Azacitidine Escalation and Expansion

SUMMARY:
This study is a first-in-human, Phase 1a/1b, multicenter, open-label study to determine the safety, tolerability, and pharmacokinetics of aplitabart as a single agent and in combination in participants with relapsed and/or refractory solid or hematologic cancers, as well as newly diagnosed cancers, and an open-label, randomized study of aplitabart+FOLFIRI+bevacizumab.

DETAILED DESCRIPTION:
Participants will be enrolled in Phase 1a, which consists of two stages: a dose-escalation stage and an expansion stage. Aplitabart will be used as a single agent and in combination with numerous other agents where standard therapeutic regimens do not exist, have proven to be ineffective or intolerable, or are considered inappropriate.

Colorectal participants may be enrolled in Phase 1b, an open-label, randomized study of aplitabart+FOLFIRI+ bevacizumab.

Aplitabart will be investigated in numerous tumor types including all-comers solid tumors, colorectal carcinoma (CRC), sarcoma, non-Hodgkin's lymphoma (NHL), acute myeloid leukemia (AML), and chronic lymphocytic leukemia (CLL).

Aplitabart will be administered intravenously (IV).

An alternative dosing schedule may be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years at time of signing ICF
* ECOG Performance Status of 0 or 1
* Histologic documentation of incurable, locally advanced or metastatic tumor of the type being evaluated in individual cohorts.
* Adequate hepatic and renal function and adequate bone marrow reserve function.
* For combination cohorts, participants must be eligible to receive the chemotherapy or targeted agent.
* Ph1a only: No more than three prior therapeutic regimens.
* Ph1b only: Must be FOLFIRI naïve participants and must have received only 1 prior therapeutic regimen administered for the treatment of cancer in the advanced/metastatic setting - OR - FOLFIRI naïve participants that only received adjuvant therapy who progressed within six months after completing adjuvant therapy, and are confirmed to have locally advanced/metastatic disease

Key Exclusion Criteria:

* Inability to comply with study and follow-up procedures.
* Prior DR5 agonist therapy.
* Concomitant use of agents well-known to cause liver toxicity.
* Concomitant use of anti-cancer agents
* Palliative radiation to bone metastases within 2 weeks prior to Day 1.
* Major surgical procedure within 4 weeks prior to Day 1.
* Untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Participants with a history of treated CNS metastases are eligible.
* Prior use of any chemotherapeutic agent or small molecule inhibitors (SMI) within 2 weeks or 5 half-lives, prior to the first dose of study treatment
* Treatment with a monoclonal antibody, or any other anticancer agent (including biologic, experimental, or hormonal therapy) investigational or otherwise, that is not chemotherapy or a SMI, within 4 weeks or five half-lives prior to first dose of study treatment.
* Ph1b: Participants who have previously received FOLFIRI treatment in the adjuvant, advanced, or metastatic disease setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Ph1a: Adverse Events of aplitabart as single agent and with FOLFIRI ± bevacizumab, aplitibart with birinapant, aplitibart with venetoclax, aplitibart with venetoclax and azacitadine, and aplitibart with gemcitabine and docetaxel | From Cycle 1 Day 1 through 28 days after the final dose of study drug
  Incidence of treatment-related AEs graded according to the NCI Common Technology Criteria for Adverse Events (CTCAE) v5.0
Ph1a: To identify the recommended expansion dose for aplitabart as single agent, with FOLFIRI ± bevacizumab, aplitibart with birinapant, aplitibart with venetoclax, aplitibart with venetoclax and azacitadine, and aplitibart with gemcitabine and docetaxel | 4 weeks
  Relationship between aplitabart dose and safety, PK, activity, and endpoints.
Ph1b: Progression-Free Survival (PFS) | Study duration of approximately 36 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 by investigator or death, whichever occurs first.

SECONDARY OUTCOMES:
Ph1a and Ph1b: Area Under the Curve (AUC) of aplitabart | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 6 months
  Area Under the Curve (AUC) of aplitabart as a single agent and in combination with the anticancer agents listed above.
Ph1a and Ph1b: Clearance (CL) of aplitabart | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 6 months
  Clearance (CL) of aplitabart as a single agent and in combination with the anticancer agents listed above.
Ph1a and Ph1b: Volume of distribution (V) of aplitabart | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 6 months
  Volume of distribution (V) of aplitabart as a single agent and in combination with the anticancer agents listed above.
Ph1a and Ph1b: Maximum Concentration (c-max) of aplitabart | At pre-defined intervals from Cycle 1 Day 1 through end of treatment at approximately 6 months
  Maximum Concentration of aplitabart as a single agent and in combination with the anticancer agents listed above.
Ph1a and Ph1b: Immunogenicity | through end of treatment at approximately 6 months
  Immunogenicity as assessed by detection of anti-drug antibodies (ADAs) to aplitabart
Ph1a and Ph1b: Objective Response Rate (ORR) | Study duration of approximately 36 months
  Preliminary efficacy of objective response rate (ORR)
Ph1a and Ph1b: Duration of Response (DoR) | Study duration of approximately 36 months
  Preliminary efficacy of duration of response (DoR)
Ph1a: Progression-Free Survival (PFS) | Study duration of approximately 36 months
  PFS is defined as the time from first dose (Ph1a) to the first documented disease progression per RECIST 1.1 by investigator or death, whichever occurs first.
Ph1a and Ph1b: Overall Survival (OS) | Study duration of approximately 36 months
  OS is defined as the time from first dose (Ph1a) or randomization (Ph1b) to death due to any cause
Ph1b: Adverse events of aplitabart + FOLFIRI + bevacizumab | From Cycle 1 Day 1 through 28 days after the final dose of study drug
  Incidence of treatment-related AEs graded according to the NCI Common Technology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Humke, MD, PhD, Study Director — IGM Biosciences
Locations (58):
- United States (37):
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Cancer and Blood Specialty Clinic (CBSC), Los Alamitos, California
  - USC Norris, Los Angeles, California
  - UCLA, Los Angeles, California
  - UC Irvine Manchester Pavilion, Orange, California
  - UCSF, San Francisco, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - SCRI at Healthone, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - FL Cancer Specialists - Lake Mary, Lake Mary, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Cancer, Jefferson, Louisiana
  - Maryland Oncology Hematology, PA - Columbia, Columbia, Maryland
  - START Midwest, Grand Rapids, Michigan
  - Minnesota Oncology - Minneapolis Clinic, Minneapolis, Minnesota
  - Mayo Clinic, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Gabrail Cancer Research, Canton, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - SCRI - Tennessee, Nashville, Tennessee
  - Texas Oncology - Austin, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - US Oncology - Dallas, Dallas, Texas
  - US Oncology- Texas Oncology - Fort Worth, Fort Worth, Texas
  - The University of Texas, MD Anderson, Houston, Texas
  - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - US Oncology- Virginia Oncology - Norfolk, Norfolk, Virginia
  - Seattle Cancer Alliance - Fred Hutch, Seattle, Washington
- Australia (6):
  - Westmead, Westmead, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Napean Cancer Care, Kingswood
  - Tasman Health, Southport
  - Queen Elizabeth Hospital, Woodville South
- France (5):
  - Institut Bergonié, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Saint Louis Hospital, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Gustave Roussy, Villejuif
- South Korea (6):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Gachon University Gil Hospital, Gyeonggi-do, Seongnam-si
  - Seoul National University Bundang Hospital, Gyeonggi-do, Seongnam-si
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital - Yonsei Cancer Center, Soeul
- Spain (4):
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Madrid FJD, Madrid
  - Madrid CIOCC - HM Universitario Sanchinnarro, Madrid

IPD SHARING:
Plan to Share IPD: No